CLINICAL TRIAL: NCT05748847
Title: Pocket Versus Tunnel Intrastromal Corneal Ring Segment Implantation (KeraRing) for the Management of Central Keratoconus
Brief Title: Pocket Versus Tunnel ICRS for Treatment of Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVTICRS
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Keratoconus
Keywords: Keratoconus; Femtosecond laser-assisted ICRS; Central keratoconus; KeraRing
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pocket ICRS (Active Comparator): Patients in this group underwent 360-degree MyoRing implantation through a femtosecond laser-assisted corneal pocket creation for the management of their central keratoconus.
  Interventions: Procedure: Intrastromal corneal ring segment implantation (Pocket)
- Tunnel ICRS (Active Comparator): Patients in this group are underwent 340-degree KeraRing implantation through a femtosecond laser-assisted corneal tunnel creation for the management of their central keratoconus.
  Interventions: Procedure: Intrastromal corneal ring segment implantation (Tunnel)

INTERVENTIONS:
Procedure: Intrastromal corneal ring segment implantation (Pocket) — Patients in this group are planned to undergo ICRS implantation through a femtosecond laser-assisted pocket creation.
  The device creates an intrastromal corneal pocket of 8-mm diameter and a depth of nearly 80% of the corneal thickness at the thinnest location with a superior tunnel incision at 90° of 5-mm width.
  Arms: Pocket ICRS
Procedure: Intrastromal corneal ring segment implantation (Tunnel) — Patients in this group are planned to undergo ICRS implantation through a femtosecond laser-assisted tunnel creation.
  The device creates an intrastromal tunnel with a depth of nearly 80% of the corneal thickness at the site of implantation. The tunnel inner and outer diameters are at 5 and 6 mm from the corneal center, respectively with the incision located at the steepest keratometry axis.
  Arms: Tunnel ICRS

SUMMARY:
Keratoconus is a corneal degenerative disease associated with loss of best-corrected visual acuity. The use of intrastromal corneal ring segment implants is indicated to regularize the cornea and to reduce aberrations.

DETAILED DESCRIPTION:
Keratoconus is a corneal degenerative disease characterized by corneal thinning and subsequent development of irregular astigmatism, diminution of vision and loss of best-corrected visual acuity.

Management of keratoconus includes halting disease progression through a corneal strengthening procedure called corneal collagen cross-linking (CXL) which usually results in stabilizing the condition but with no improvement in visual acuity or quality. Intrastromal corneal ring segment (ICRS) implantation is a well-established procedure for the management of moderate keratoconus with a corneal flattening effect that is associated with improvement of visual acuity and reduction of optical aberrations.

The aim of the study is to evaluate and compare the visual, refractive and topographic outcomes of two different femtosecond laser assisted surgical techniques to create a corneal stromal pocket or a tunnel for implantation of ICRS for the management of central keratoconus

ELIGIBILITY:
Inclusion Criteria:

1. Patients with progressive keratoconus with maximum keratometry (Kmax) between 50-65 diopters
2. Central keratoconus (Keratoconus with steepest corneal point within the central 3 mm zone).
3. Clear corneal with a minimum pachymetry of 400 μm.

Exclusion Criteria:

1. Corneal scars
2. Patients with advanced keratoconus with Kmax > 65 diopters.
3. Non-central keratoconus (para-central or peripheral keratoconus with steepest corneal point outside the central 3 mm zone).
4. Previous corneal cross-linking and/or ocular surgery.
5. Systemic diseases such as diabetes mellitus and autoimmune diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Complications | 12 months
  Postoperative complications following intrastromal corneal ring segment implantation.
Postoperative keratometry | 12 months
  Postoperative keratometry as measured by Scheimpflug imaging Pentacam
Postoperative Refraction | 12 months
  Spherical equivalent refraction measured by Topcon Auto-Keratorefractometer
Corrected distance visual acuity (CDVA) | 12 months
  Corrected distance visual acuity measurement using Snellen's Acuity Chart expressed as logMAR notation
Uncorrected distance visual acuity (UDVA) | 12 months
  Uncorrected distance visual acuity measurement using Snellen's Acuity Chart expressed as logMAR notation

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, MD, Principal Investigator — Assiut University
Locations (1):
- Tiba Eye Center, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Izquierdo L Jr, Rodriguez AM, Sarquis RA, Altamirano D, Henriquez MA. Intracorneal circular ring implant with femtosecond laser: Pocket versus tunnel. Eur J Ophthalmol. 2022 Jan;32(1):176-182. doi: 10.1177/1120672121994729. Epub 2021 Feb 12. PMID 33579160
- [Derived] Abdel-Radi M, Anwar M, Mostafa MM. Complications and Outcomes of Femtosecond Laser-Assisted Corneal Pocket Implantation of 360-Degree MyoRing(R) Versus Corneal Tunnel Implantation of 340-Degree Keraring(R) for the Management of Central Keratoconus. Curr Eye Res. 2025 Nov 20:1-9. doi: 10.1080/02713683.2025.2587890. Online ahead of print. PMID 41263332